CLINICAL TRIAL: NCT04536961
Title: A Phase 1, Open-label, Crossover Study to Evaluate the Pharmacokinetics of BMS-986165 Administered as Various Prototypic Solid Tablet Formulations in Healthy Subjects
Brief Title: A Study to Evaluate the Drug Levels of BMS-986165 When Taken as Various Solid Tablet Prototypes by Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-136
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers
MeSH Terms: interventions — deucravacitinib; Famotidine; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Part A: Reference Treatment (Experimental)
  Interventions: Drug: Reference Treatment- BMS-986165-01
- Part A Prototype (Experimental)
  Interventions: Drug: Prototype BMS-986165
- Part C Reference Treatment (Experimental)
  Interventions: Drug: Reference Treatment- BMS-986165-01
- Part C: Prototype (Experimental)
  Interventions: Drug: Prototype BMS-986165
- Part B: Treatment 1 (Experimental)
  Interventions: Drug: Prototype BMS-986165
- Part B: Treatment 2 (Experimental)
  Interventions: Drug: Prototype BMS-986165
- Part B: Treatment 3 (Experimental)
  Interventions: Drug: Prototype BMS-986165
- Part B: Treatment 4 (Experimental)
  Interventions: Drug: Prototype BMS-986165; Drug: Famotidine
- Part B: Treatment 5 (Experimental)
  Interventions: Drug: Prototype BMS-986165; Other: Alcohol

INTERVENTIONS:
Drug: Reference Treatment- BMS-986165-01 — Specified dose on specified days
  Other Names: Deucravacitinib
  Arms: Part A: Reference Treatment; Part C Reference Treatment
Drug: Prototype BMS-986165 — Specified dose on specified days
  Other Names: Deucravacitinib
  Arms: Part A Prototype; Part B: Treatment 1; Part B: Treatment 2; Part B: Treatment 3; Part B: Treatment 4; Part B: Treatment 5; Part C: Prototype
Drug: Famotidine — Specified dose on specified days
  Arms: Part B: Treatment 4
Other: Alcohol — Specified quantity on specified days
  Arms: Part B: Treatment 5

SUMMARY:
The purpose of this study is to evaluate the drug levels of BMS-986165 in when taken by mouth as various solid tablet prototypes, by healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* No clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations.
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive, and total body weight ≥50 kg (110 lb). BMI = weight (kg)/(height [m])2 at screening.
* Willing and able to consume 4 units of alcohol (Part B only)
* A negative polymerase chain reaction (PCR) test for coronavirus disease 2019 (COVID-19) at screening and admission
* Males and females must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Current or recent (within 3 months or 90 days of study drug administration) clinically significant gastrointestinal disease that, in the opinion of the investigator or medical monitor, could impact upon the absorption of study drug
* Any medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of or active liver disease.
* Clinically significant history or presence of acute or chronic bacterial, fungal, or viral infection (eg, pneumonia, septicemia) within the 3 months or 90 days prior to screening.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986165 | Day 1 and Day 7
Time of maximum observed plasma concentration (Tmax) of BMS-986165 | Day 1 and Day 7
Area under the plasma concentration-time curve from time zero to t (AUC (0-t)) of BMS-986165 | Day 1 and Day 7
  Part A, B, C

SECONDARY OUTCOMES:
Incidence of Nonserious Adverse Events (AEs) | Up to approximately 60 days (for Parts A & C), approximately 69 days (for Part B)
Incidence of Serious Adverse Events (AEs) | Up to approximately 83 days (for Parts A & C), approximately 92 days (for Part B)
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
Incidence of clinically significant changes in vital signs: Blood pressure | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
Incidence of clinically significant changes in vital signs: Heart rate | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
Incidence of clinically significant changes in vital signs: Body temperature | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave.
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
  The QT interval is the time from the start of the Q wave to the end of the T wave.
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to approximately 53 days (for Parts A & C), approximately 62 days (for Part B)
  PR interval is the time from the onset of the P wave to the start of the QRS complex

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Quotient Sciences Miami, Nottingham, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm